CLINICAL TRIAL: NCT03751332
Title: The Vienna Prograf and Endothelial Progenitor Cell Extension Study
Acronym: PEP-X
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gere Sunder-Plassmann, Associated Professor of Medicine, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.05; 154/01/2008 (Other: Ethics Committee Medical University of Vienna)
Record Dates: First submitted 2018-11-09; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Immunosuppression; Renal Failure
Keywords: Calcineurin inhibitors; Tacrolimus modified release; Conversion; Trough levels; MDR-1
MeSH Terms: conditions — Renal Insufficiency | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conversion from either CSA or TAC (Other): Tacrolimus with modified galenic (tacrolimus MR4; Advagraf®) once daily. In patients treated with ciclosporin A, the initial dose will be 0.1 - 0.12 mg tacrolimus MR4 per kg of body weight per day with oral morning administration. In patients who are already treated with Prograf, the conversion to Advagraf will be performed in a 1:1 ratio.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Conversion from either cyclosporin or tacrolimus to tacrolimus modified release

SUMMARY:
Conversion of renal transplant recipients from either tacrolimus or cyclosporin A to tacrolimus modified release to investigate the effects of the MDR1/CYP450 genotype on the trough blood levels of tacrolimus with modified galenic (tacrolimus MR4; Advagraf®).

DETAILED DESCRIPTION:
The study concerns the conversion of immunosuppressive agents among participants in the clinical trial "The Vienna Prograf and Endothelial Progenitor Cell Study - The Vienna PEP Study" at the end of the study after 2 years in the extension study PEP-X.

The aim of the conversion is to investigate the effects of the multi-drug resistance (MDR1, gene symbol ABCB1) genotype on the trough blood levels of tacrolimus modified release (TAC MR4; Advagraf®). Analyzes of the effects of the genotype on the concentration/dose ratio ([ng/mL]/[mg/d]) will be carried out, as well as studies on existing polymorphisms in the MDR1 gene. The written informed consent to conversion of either tacrolimus (TAC; Prograf®) or cyclosporin A (CSA; Sandimmun Neoral®) to TAC MR4 will be obtained.

Upon completion of 24 months of study participation of the PEP-study, and consent to convert the immunosuppressant therapy of either TAC or CSA to TAC MR4, it will be used as indicated by the manufacturer. In patients treated with CSA, the initial dose will be 0.1-0.12 mg TAC MR4 per kg of body weight per day with oral morning administration. In patients who are already treated with TAC, the conversion to TAC MR4 will be performed in a 1:1 ratio.

The dosage data for the conversion of CSA to TAC MR4 are taken from the documents of the European Medicines Agency homepage (http://www.emea.europa.eu/index/ indexh1.htm, retrieved 26.09.2007), those on the safety and equivalence of the achieved areas under the curve (AUC) of both TAC formulations from Alloway et al. (Transplant Proc 2005; 37: 867-870).

The conversion will be performed by Univ. Prof. Dr. Gere Sunder-Plassmann, and Dr. Markus Riegersperger, respectively, both Division of Nephrology and Dialysis, Department of Medicine III, Medical University of Vienna, Währinger Gürtel 18-20, 1090 Vienna. The desired trough level is set at 4.0-8.0ng/mL according to the usual clinical standards for long-term transplant patients at the investigators center. The trough level analyses are performed at the Medical University of Vienna, according to the following schedule: 1 week after conversion, 2 weeks after conversion, 4 weeks after conversion, 12 weeks and 12 months after conversion.

ELIGIBILITY:
Inclusion Criteria:

* Any stable long-term kidney transplant recipient who participated in the Vienna Prograf and Endothelial-Progenitor Study (Vienna PEP Study; EudraCT identifier 2004-82 004209-98)
* Written informed consent to have the immunosuppression converted from either cyclosporin A or tacrolimus to tacrolimus modified-release

Exclusion Criteria:

* Graft failure
* Contraindication to receive immunosuppression

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Effects of the MDR1 genotype on the trough blood levels of tacrolimus with modified galenics (tacrolimus MR4; Advagraf®) | 12 months
  Effects of the genotype on the concentration/dose ratio ([ng/mL]/[mg/d])

CONTACTS AND LOCATIONS:
Overall Officials: Gere Sunder-Plassmann, MD, Principal Investigator — Medical University of Vienna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Riegersperger M, Plischke M, Jallitsch-Halper A, Steinhauser C, Fodinger M, Winkelmayer WC, Dunkler D, Sunder-Plassmann G. A non-randomized trial of conversion from ciclosporin and tacrolimus to tacrolimus MR4 in stable long-term kidney transplant recipients: Graft function and influences of ABCB1 genotypes. PLoS One. 2019 Jul 2;14(7):e0218709. doi: 10.1371/journal.pone.0218709. eCollection 2019. PMID 31266056